CLINICAL TRIAL: NCT06082817
Title: An Open-Label Pilot Study of the Pharmacokinetics and Safety of 50 Mg Oral Testosterone Undecanoate (Kyzatrex) in Menopausal Women with Low Testosterone and Hypoactive Sexual Desire Disorder
Brief Title: An Open-Label Study of 50 Mg Oral Testosterone Undecanoate (Kyztrex) in Menopausal Women with Low Testosterone and HSDD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego Sexual Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDSM-2023-03
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Hypoactive Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Open label 50mg daily dosing with pharmacokinetics assessed by multiple blood draws
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): Participants will receive 50mg oral testosterone undecanoate daily, have pharmacokinetics assessed and complete validated instruments
  Interventions: Drug: Oral Testosterone Undecanoate

INTERVENTIONS:
Drug: Oral Testosterone Undecanoate — 50mg oral testosterone undecanoate daily
  Other Names: Kyzatrex

SUMMARY:
This is an unblinded study to be conducted at a single research center, San Diego Sexual Medicine. Eligible subjects will receive 50 mg capsules of Kyzatrax® to be taken orally daily over a 3-month period. Multiple blood samples will be taken at baseline and on days 7, 28 and 56 to assess safety and pharmacokinetics of the testosterone. After the informed consent is signed and for up to 14 days after the last dose of study drug, participants will have serial blood samples collected in addition to other routine study procedures (e.g. vital signs measured, adverse events assessed, validated outcome scales completed).

DETAILED DESCRIPTION:
This study is being conducted in an unblinded fashion because the primary endpoint is pharmacokinetic information, and all subjects will receive the same active drug at the same dosage. The primary objectives of this study are to assess the short-term safety and to investigate the pharmacokinetics of serum concentration of total testosterone with daily administration of one (1) 50 mg capsule of testosterone undecanoate (Kyzatrax®) in thirty menopausal women with hypoactive sexual desire disorder (HSDD) and low testosterone. The secondary objective of this study is to assess the efficacy of daily oral administration of one (1) 50 mg capsule of testosterone undecanoate (Kyzatrax®) in thirty menopausal women with HSDD and low testosterone.

The eligibility criterion for testosterone concentration (< 25 ng/mL [< 0.87 nmol/L]) is based on the lower limit of the normal testosterone reference range for adult females. The dose of 50 mg was chosen because this is the lowest oral testosterone currently being manufactured and it represents 12.5% of the starting dose of Kyzatrex FDA approved for men (see Attachment 1). Based on the guidelines of the International Society for the Study of Women's Sexual Health, the starting dose of testosterone for peri- and post-menopausal women is approximately 10% of a testosterone product FDA approved for men. In clinical practice, women are typically prescribed testosterone therapy at 10-20% of the dose given to men, depending on individual adsorption and metabolism characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Participant provides written informed consent and HIPAA authorization before any study procedures are conducted;
2. Participant is female;
3. Participant is aged 30 years or greater;
4. Participant is menopausal either spontaneously (at least 12 months amenorrheic or 6 months amenorrheic and FSH >40 IU/ml) or 6 weeks after bilateral salpingo-oophorectomy with or without hysterectomy.
5. Participant has a body mass index (BMI) ≤ 34 kg/m2;
6. Participant has a diagnosis of hypoactive sexual desire disorder;
7. At screening, participant has a testosterone concentration <30 ng/dL;
8. Participant has a normal PAP smear within 6 months of first administration of study drug if participant has a cervix;
9. Participant has a normal mammogram within 6 months of first administration of study drug;
10. Participant agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Participant has a hypersensitivity to testosterone, gelatin, glycerin, sorbitol, or titanium dioxide (the constituents of Kyzatrex capsule);
2. Participant has received intramuscular testosterone injections, oral or transdermal testosterone within 4 weeks, or subcutaneous testosterone pellet within 6 months prior to the screening visit, or receives any form of testosterone other than study drug during this trial;
3. Participant has documented or suspected breast cancer, history of heart attack or stroke;
4. Participant has a clinically significant history of disease which could alter absorption, distribution, metabolism, or elimination, such as hepatic, renal, hematologic, gastrointestinal, respiratory, endocrine, or neurological disease;
5. Participant has an EKG with an abnormality of clinical significance;
6. Participant has an abnormal PAP smear if she has a cervix;
7. Participant has any chronic medical condition or psychologic disorder that the Principal Investigator feels makes her ineligible for the study;
8. Participant requires major surgery within 4 weeks before signing consent or at any time during the study;
9. Participant requires a treatment with any medication listed in Appendix 1 at any time between 30 days before study drug is started or any time until the end of the study;
10. Participant has a history of substance abuse within 12 months prior to signing consent;
11. Participant has received an investigational drug within 30 days prior to signing consent;
12. Participant has any condition or exhibits behavior that indicates to the Principal Investigator that the participant is unlikely to be compliant with study procedures and visits.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender female identifying as a female
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Testosterone | days 0, 7, 28, 56
  serum concentration of total testosterone to assess safety (adverse events) and pharmacokinetics

SECONDARY OUTCOMES:
Female Sexual Function Index | Days 0, 28, 56, 84
  Female Sexual Function Index to assess changes in each domain and total, total range 2-36, lower the score the more dysfunction therefore worse function

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clayton AH, Goldstein I, Kim NN, Althof SE, Faubion SS, Faught BM, Parish SJ, Simon JA, Vignozzi L, Christiansen K, Davis SR, Freedman MA, Kingsberg SA, Kirana PS, Larkin L, McCabe M, Sadovsky R. The International Society for the Study of Women's Sexual Health Process of Care for Management of Hypoactive Sexual Desire Disorder in Women. Mayo Clin Proc. 2018 Apr;93(4):467-487. doi: 10.1016/j.mayocp.2017.11.002. Epub 2018 Mar 12. PMID 29545008
- [Background] Parish SJ, Simon JA, Davis SR, Giraldi A, Goldstein I, Goldstein SW, Kim NN, Kingsberg SA, Morgentaler A, Nappi RE, Park K, Stuenkel CA, Traish AM, Vignozzi L. International Society for the Study of Women's Sexual Health Clinical Practice Guideline for the Use of Systemic Testosterone for Hypoactive Sexual Desire Disorder in Women. J Sex Med. 2021 May;18(5):849-867. doi: 10.1016/j.jsxm.2020.10.009. Epub 2021 Apr 1. PMID 33814355
- [Background] Bachmann G, Bancroft J, Braunstein G, Burger H, Davis S, Dennerstein L, Goldstein I, Guay A, Leiblum S, Lobo R, Notelovitz M, Rosen R, Sarrel P, Sherwin B, Simon J, Simpson E, Shifren J, Spark R, Traish A; Princeton. Female androgen insufficiency: the Princeton consensus statement on definition, classification, and assessment. Fertil Steril. 2002 Apr;77(4):660-5. doi: 10.1016/s0015-0282(02)02969-2. PMID 11937111
- [Background] Davis SR, Wahlin-Jacobsen S. Testosterone in women--the clinical significance. Lancet Diabetes Endocrinol. 2015 Dec;3(12):980-92. doi: 10.1016/S2213-8587(15)00284-3. Epub 2015 Sep 7. PMID 26358173
- [Background] White WB, Bernstein JS, Rittmaster R, Dhingra O. Effects of the oral testosterone undecanoate Kyzatrex on ambulatory blood pressure in hypogonadal men. J Clin Hypertens (Greenwich). 2021 Jul;23(7):1420-1430. doi: 10.1111/jch.14297. Epub 2021 Jun 11. PMID 34114726
- [Background] Asghar AA, Hashmi MR, Ahmed R, Khabir Y. Kyzatrex - Oral testosterone replacement therapy. Ann Med Surg (Lond). 2022 Sep 11;82:104625. doi: 10.1016/j.amsu.2022.104625. eCollection 2022 Oct. No abstract available. PMID 36268410